CLINICAL TRIAL: NCT00888433
Title: Renal Denervation in Patients With Uncontrolled Hypertension (Symplicity HTN-2)
Acronym: HTN-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Vascular (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: TP-058
Record Dates: First submitted 2009-04-24; First posted 2009-04-27 (Estimated); Results first posted 2014-02-24 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2015-05

CONDITIONS: Uncontrolled Hypertension
Keywords: hypertension; renal denervation; sympathetic nervous system; RDN
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Renal Denervation (Experimental): Renal Denervation and maintenance of anti-hypertensive medications
  Interventions: Device: Renal Denervation (Symplicity® Renal Denervation System)
- Control (No Intervention): Maintenance of anti-hypertensive medications with option for cross-over treatment after 6-months

INTERVENTIONS:
Device: Renal Denervation (Symplicity® Renal Denervation System) — Catheter-based renal denervation
  Arms: Renal Denervation

SUMMARY:
An international, multi-center, prospective, randomized, controlled study of the safety and effectiveness of renal denervation in patients with uncontrolled hypertension.

ELIGIBILITY:
Inclusion Criteria:

* systolic blood pressure >=160mmHg (>=150 mmHg for type 2 diabetics);
* on 3 or more antihypertensive medications
* >= 18 and =< 85 years of age.

Exclusion Criteria:

* renal artery abnormalities
* eGFR < 45mL/min
* MI, angina, CVA within 6 months
* Type 1 diabetes
* ICD or pacemaker, or any other metallic implant not compatible with MRI
* others

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2009-06; Primary Completion 2010-09 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Murray Esler, MBBS, Principal Investigator — The Baker IDI Heart & Diabetes Institute
Locations (20):
- Alfred Hospital, Melbourne, Australia
- Vienna General Hospital, Vienna, Austria
- Cliniques Universitaires Saint Luc, Brussels, Belgium
- Hopital Européen Georges Pompidou, Paris, France
- Germany (9):
  - Herzzentrum Bad Krozingen, Bad Krozingen
  - Universität zu Köln, Cologne
  - Universitaetsklinikum Dusseldorf, Düsseldorf
  - University of Erlangen at Nuremburg, Erlangen
  - Universitaetsklinikum Essen, Essen
  - CardioVascular Center Frankfurt, Frankfurt
  - Universitatskliniken des Saarlandes, Homburg
  - University of Leipzig - Herzzentrum, Leipzig
  - Universitatsklinikum Schleswig-Holstein, Luebeck Campus, Leubeck
- Pauls Stradins Clinical University Hospital, Riga, Latvia
- Samodzielna Pracownia Hemodynamiczna, Warsaw, Poland
- Hospital 12 de Octubre, Madrid, Spain
- Universitaatsspital Zurich, Zurich, Switzerland
- United Kingdom (3):
  - Kent and Canterbury Hospital, Canterbury
  - University of Glasgow, Glasgow
  - Barts and the London School of Dentistry & Medicine, London

REFERENCES:
- [Result] Symplicity HTN-2 Investigators; Esler MD, Krum H, Sobotka PA, Schlaich MP, Schmieder RE, Bohm M. Renal sympathetic denervation in patients with treatment-resistant hypertension (The Symplicity HTN-2 Trial): a randomised controlled trial. Lancet. 2010 Dec 4;376(9756):1903-9. doi: 10.1016/S0140-6736(10)62039-9. Epub 2010 Nov 17. PMID 21093036
- [Derived] Eikelis N, Hering D, Marusic P, Duval J, Hammond LJ, Walton AS, Lambert EA, Esler MD, Lambert GW, Schlaich MP. The Effect of Renal Denervation on Plasma Adipokine Profile in Patients with Treatment Resistant Hypertension. Front Physiol. 2017 May 30;8:369. doi: 10.3389/fphys.2017.00369. eCollection 2017. PMID 28611687
- [Derived] Schmieder RE, Ott C, Schmid A, Friedrich S, Kistner I, Ditting T, Veelken R, Uder M, Toennes SW. Adherence to Antihypertensive Medication in Treatment-Resistant Hypertension Undergoing Renal Denervation. J Am Heart Assoc. 2016 Feb 12;5(2):e002343. doi: 10.1161/JAHA.115.002343. PMID 26873693
- [Derived] Esler MD, Bohm M, Sievert H, Rump CL, Schmieder RE, Krum H, Mahfoud F, Schlaich MP. Catheter-based renal denervation for treatment of patients with treatment-resistant hypertension: 36 month results from the SYMPLICITY HTN-2 randomized clinical trial. Eur Heart J. 2014 Jul;35(26):1752-9. doi: 10.1093/eurheartj/ehu209. Epub 2014 Jun 4. PMID 24898552
- [Derived] Mahfoud F, Ukena C, Schmieder RE, Cremers B, Rump LC, Vonend O, Weil J, Schmidt M, Hoppe UC, Zeller T, Bauer A, Ott C, Blessing E, Sobotka PA, Krum H, Schlaich M, Esler M, Bohm M. Ambulatory blood pressure changes after renal sympathetic denervation in patients with resistant hypertension. Circulation. 2013 Jul 9;128(2):132-40. doi: 10.1161/CIRCULATIONAHA.112.000949. Epub 2013 Jun 18. PMID 23780578
- [Derived] Esler MD, Krum H, Schlaich M, Schmieder RE, Bohm M, Sobotka PA; Symplicity HTN-2 Investigators. Renal sympathetic denervation for treatment of drug-resistant hypertension: one-year results from the Symplicity HTN-2 randomized, controlled trial. Circulation. 2012 Dec 18;126(25):2976-82. doi: 10.1161/CIRCULATIONAHA.112.130880. PMID 23248063
- [Derived] Ukena C, Mahfoud F, Kindermann I, Barth C, Lenski M, Kindermann M, Brandt MC, Hoppe UC, Krum H, Esler M, Sobotka PA, Bohm M. Cardiorespiratory response to exercise after renal sympathetic denervation in patients with resistant hypertension. J Am Coll Cardiol. 2011 Sep 6;58(11):1176-82. doi: 10.1016/j.jacc.2011.05.036. PMID 21884958
- [Derived] Mahfoud F, Schlaich M, Kindermann I, Ukena C, Cremers B, Brandt MC, Hoppe UC, Vonend O, Rump LC, Sobotka PA, Krum H, Esler M, Bohm M. Effect of renal sympathetic denervation on glucose metabolism in patients with resistant hypertension: a pilot study. Circulation. 2011 May 10;123(18):1940-6. doi: 10.1161/CIRCULATIONAHA.110.991869. Epub 2011 Apr 25. PMID 21518978
- [Derived] Schlaich MP, Straznicky N, Grima M, Ika-Sari C, Dawood T, Mahfoud F, Lambert E, Chopra R, Socratous F, Hennebry S, Eikelis N, Bohm M, Krum H, Lambert G, Esler MD, Sobotka PA. Renal denervation: a potential new treatment modality for polycystic ovary syndrome? J Hypertens. 2011 May;29(5):991-6. doi: 10.1097/HJH.0b013e328344db3a. PMID 21358414
- See also: Related Info — http://www.medtronicrdn.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 190 patients screened as eligible for study inclusion between June 9, 2009 and January 15, 2010.
Pre-assignment Details: 84 subjects excluded pre-randomization due to blood pressure value at baseline visit (n=36); ineligible anatomy (n=30); declined participation (n=10); and other exclusion criteria (n=8).
Period: Overall Study
Arm/Group | Renal Denervation | Control
Started | 52 | 54
Completed | 49 | 51
Not Completed | 3 | 3
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Missed Visit | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Renal Denervation | Control | Total
Number analyzed (Participants) | 52 | 54 | 106
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.2 (11.9) | 58.3 (12.3) | 58.2 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 27 | 45
  Male | 34 | 27 | 61
Region of Enrollment [Number; unit: participants]
  France | 1 | 3 | 4
  Poland | 1 | 1 | 2
  Belgium | 4 | 2 | 6
  Spain | 2 | 2 | 4
  Australia | 5 | 5 | 10
  Austria | 1 | 2 | 3
  Latvia | 3 | 4 | 7
  Germany | 32 | 29 | 61
  Switzerland | 0 | 1 | 1
  United Kingdom | 3 | 5 | 8

OUTCOME MEASURES:

1. Primary Outcome: Office Systolic Blood Pressure Reduction
Description: The primary effectiveness endpoint is change in Office Systolic Blood Pressure (SBP) from baseline to 6 months post-randomization.
Time Frame: Baseline to 6 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Renal Denervation | Control
Number analyzed (Participants) | 49 | 51
mmHg | -31.7 (23.1) | 0.9 (20.6)

ADVERSE EVENTS:
Time Frame: 12 months
Groups:
- 1. DENERVATION: Renal Denervation and maintenance of anti-hypertensive medications
- 2. CONTROL: Maintenance of anti-hypertensive medications with option for cross-over treatment after 6-months
Arm/Group | 1. DENERVATION | 2. CONTROL
Serious Adverse Events (participants affected / at risk) | 5/52 | 4/54
Other Adverse Events (participants affected / at risk) | 18/52 | 7/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1. DENERVATION (N=52) | 2. CONTROL (N=54)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0)
Oedema (General disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Cerebrovascular Accident (Nervous system disorders) | 0 (0) | 1 (1)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0)
Intra-Cerebral Aneurysm Operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (2) | 1 (1)
Hypertensive Crisis (Vascular disorders) | 2 (2) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1. DENERVATION (N=52) | 2. CONTROL (N=54)
Bradycardia (Cardiac disorders) | 3 (3) | 0 (0)
Oedema Peripheral (General disorders) | 3 (6) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 5 (13) | 0 (0)
Dizziness (Nervous system disorders) | 4 (6) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 3 (7)
Hypertensive Crisis (Vascular disorders) | 0 (0) | 4 (7)
Hypotension (Vascular disorders) | 3 (5) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The institution agrees that no Publication of the Study Results may be made until Publication of the results of the multi-centre study or 2 years after Study Completion, whichever is sooner.